CLINICAL TRIAL: NCT05289232
Title: Prevalence of Complications Post Sutured Wounds in the ED
Brief Title: Prevalence and Complications of Suture in the ED
Status: Completed | Type: Observational
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, Professor, University of Monastir
Other Study IDs: suture
Record Dates: First submitted 2022-03-02; First posted 2022-03-21 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Suture, Complication
Keywords: suture; complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
included patients who had sutured wounds in the ED were asked about complications after suture .

DETAILED DESCRIPTION:
All patients using the emergency room of EPS Fattouma Bourguiba Monastir are welcomed by a resident in the suture room. After an inclusion, patients are cared for in the outpatient circuit and the suture will be done in the dedicated box. Before discharging the patient, instructions and standardized prescriptions are given to the patient such as standard prescriptions for local wound care, removal of stitches and verification of vaccination status.

The data relevant to this study are obtained prospectively from a detailed questionnaire in the annex and a telephone call and they are completed retrospectively with the data collected in the computerized medical record.

At the healing period, between 15 days and 45 days after the suture, the investigators called the patients back in order to know the evolution of the wound, the adherence to the instructions and the prescriptions, the quality of healing and the search for complications (infection , loose stitches, hematoma, etc.)

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute suturable wound

Exclusion Criteria:

Wounds requiring surgical treatment Septic wounds Chronic lesions Vascular wounds Patients who did not consent to the protocol.

Ages: 12 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Included patients presented to the outpatient emergency circuit of the EPS Fattouma Bourguiba Monastir having as main reason for consultation an acute suturable wound. The patients excluded are those who consulted for wounds requiring surgical treatment, septic wounds and patients who did not consent to the protocol.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Sutures complications after discharge of the Emergency Department PART 1 | 15 days after the suture
  After discharge from ED , patients were called back in order to know other informations about the patient and about the wound : its location,its dimension,the edges of the wound ,if its bleedong before suture ,and other factors that can facilitate its complications . the evolution of the wound, the adherence to the instructions and the prescriptions, the quality of healing and the search for complications

SECONDARY OUTCOMES:
Sutures complications after discharge of the Emergency Department PART 2 | 45 days after the suture
  the patients were asked about the evolution of the wound,the appearence of complications such as disunity of stitches ,infection,delayed healing, necrosis, subcutaneous hematoma and about the adherence to the instructions and the prescriptionsgiven at discharge .

CONTACTS AND LOCATIONS:
Overall Officials: Semir Nouira, Professor, Principal Investigator — University of Monastir
Locations (1):
- Emergency department of university hospital Fattouma Bourguiba of Monastir Monastir, Monastir Tunisia Monastir, Tunisia, 5000, Monastir, Monastir ,Tunisia, Tunisia